CLINICAL TRIAL: NCT00427700
Title: Induction of Ovulation With Raloxifene or Clomiphene Citrate in Polycystic Ovarian Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RACLO
Record Dates: First submitted 2007-01-26; First posted 2007-01-29 (Estimated); Results first posted 2016-10-06 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2024-07

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome; clomiphene citrate; Raloxifene
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Clomiphene; Raloxifene Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clomiphene (Active Comparator): Uso of 100mg of clomiphene citrate during days 5-9 of the menstrual cycle
  Interventions: Drug: clomiphene citrate
- Raloxifene (Experimental): Use of 100mg of raloxifene during days 5-9 of the menstrual cycle
  Interventions: Drug: raloxifene

INTERVENTIONS:
Drug: clomiphene citrate — 100mg PO on days 5-9 of the menstrual cycle
  Other Names: Clomid
  Arms: Clomiphene
Drug: raloxifene — 100mg PO on days 5-9 of the menstrual cycle
  Other Names: Evista
  Arms: Raloxifene

SUMMARY:
The Polycystic Ovarian Syndrome (PCOS) is a common disorder related to ovulation problems. Clomiphene citrate (CC) is the drug of first choice for this condition. Nevertheless, CC has a detrimental effect over uterine receptivity.

Raloxifene is a Selective Estrogen Receptor Modulator, that does not have a detrimental effect over the endometrium, and also increase the serum levels of FSH, thus, inducting ovulation.

The objective of this study is to compare the ovulation rate in PCOS patients between clomiphene citrate and raloxifene in a double blind randomized trial.

DETAILED DESCRIPTION:
-Introduction The Polycystic Ovarian Syndrome (PCOS) is a frequent endocrine among women in reproductive ages, with a prevalence of 10%. In 2003, a consensus among the European and American Society of Human Reproduction (ESRHE and ASRM) defined that PCOS is a ovarian disfunction which present at least 2 out of 3 criteria: oligomenorrhea or anovulation; clinical or laboratorial signs of hyperandrogenism and polycystic ovaries on ultrasound; other causes, such as congenital adrenal hyperplasia, androgen secretory tumors, Cushing syndrome and hyperprolactinemia must be rule out.

Patients with PCOS who desire to became pregnant need, in their majority, induction of ovulation. Traditionally, clomiphene citrate, an estrogen receptor agonist, is the most used drug for this type of anovulation. The mechanism of action of clomiphene is related to a negative feedback to the endogenous estrogen, resulting in a higher amplitude of gonadotrophin surges, i.e., luteinizing hormone(LH) and follicle stimulating hormone(FSH). Nevertheless, recent studies have been shown that clomiphene citrate has a deleterious effect in the endometrium. The markers of uterine receptivity, among them, the integrin beta3 subunit, has its expression diminished, which implicate in a reduced fecundation rate.

The raloxifene is a selective estrogen receptor modulator. It has an agonist and antagonist activity over different organs. The daily therapy with raloxifene increase bone density, reduce cholesterol serum concentrations (LDL) and do not stimulate the endometrium in post-menopausal women (Delmas PD et al., 1997). Recent studies have shown that this drug is safe in healthy pre-menopausal women (Baker VL et al., 1998). A daily dosi of 100mg per 28 days, beginning on the 3rd day of the cycle, has shown that FSH and LH levels were not affected when compared to controls during the menstrual cycle. However, women who had received 100mg of raloxifene had a 31% increase in their FSH serum levels during the follicular phase, when compared to controls. An increase to 200mg did not increase FSH levels (Baker VL et al, 1998). Furthermore, it has been shown that raloxifene significantly increase the in vitro expression of αvβ3 integrin, suggesting a beneficial effect over the endometrium in relation to clomiphene (Lessey BA, personal communication, 2006).

-Objective To compare the ovulation rate between raloxifene and clomiphene among women with polycystic ovarian syndrome.

To identify the endometrial alterations compatible with ovulations, i.e., secretory endometrium, through endometrial biopsy between the women who used raloxifene or clomiphene.

-Patients and Methods

Patients with the diagnosis of polycystic ovarian syndrome (because of infertility or hirsutism) who had a consultation at outpatient clinic of Hospital de Clínicas de Porto Alegre will be invited to participate in the study, after signing the informed consent. A standard interview will be performed. In the first consultation, the laboratorial exams will reviewed: total testosterone, 17 OH-progesterone, fasting glucose, TSH, prolactin. After the interview, the patient will be randomized for one of the treatments:

100mg of clomiphene or 100mg of raloxifene from day 3 of the menstrual cycle, for 5 days. Menstruation will be induced with 10mg of oral medroxyprogesterone per 10 days. On day 10, urinary LH will be collected daily along with endovaginal ultrasound for assessing follicular development. On post-ovulatory day 8~10, progesterone levels will be measured from blood. An endometrial biopsy on day 8~10 post-ovulation will be performed in those patients who do not wish to became pregnant. The endometrial biopsy will divided into 2 parts and kept in liquid nitrogen and formol for immunohistochemistry and histological analysis respectively.

Sample size and statistical analysis

Ethical aspects

ELIGIBILITY:
Inclusion Criteria:

* All patients with polycystic ovarian syndrome will be invited to participate in the study. The PCOS criteria are according to modified Rotterdam criteria (7); i.e., oligoovulation defined as < 6 menstrual periods per year, signs of clinical hyperandrogenism (Ferriman and Gallwey >8) or laboratorial (total Testosterone >=0.81 ng/dL) or polycystic ovary > 10cm3.

Furthermore, all patients with infertility diagnosis based solely on ovulation factor will included in the protocol

* Age >18 years old and <= 38 years old.
* No endometriosis on laparoscopy

Exclusion Criteria:

* Not willing to participate in the study
* use of IUD or contraceptive pill within 2 months before the study.
* Hyperprolactinemia (>20ng/mL)
* Abnormal serum levels of TSH(normal range:0.4-40 mUI/mL).
* High 17-OH progesterone (>=4.9ng/mL)
* Endometriosis
* Known allergy to clomiphene or raloxifene

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2008-08; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo F Savaris, MD, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre; Helena Corleta, MD, PhD, Study Chair — Hospital de Clínicas de Porto Alegre; Bruce A Lessey, MD, PhD, Study Director — Greenville Hospital System
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Delmas PD, Bjarnason NH, Mitlak BH, Ravoux AC, Shah AS, Huster WJ, Draper M, Christiansen C. Effects of raloxifene on bone mineral density, serum cholesterol concentrations, and uterine endometrium in postmenopausal women. N Engl J Med. 1997 Dec 4;337(23):1641-7. doi: 10.1056/NEJM199712043372301. PMID 9385122
- [Background] Baker VL, Draper M, Paul S, Allerheiligen S, Glant M, Shifren J, Jaffe RB. Reproductive endocrine and endometrial effects of raloxifene hydrochloride, a selective estrogen receptor modulator, in women with regular menstrual cycles. J Clin Endocrinol Metab. 1998 Jan;83(1):6-13. doi: 10.1210/jcem.83.1.4448. PMID 9435408
- [Background] Grimes DA. The "CONSORT" guidelines for randomized controlled trials in Obstetrics & Gynecology. Obstet Gynecol. 2002 Oct;100(4):631-2. doi: 10.1016/s0029-7844(02)02233-0. No abstract available. PMID 12383524
- [Background] Moher D, Schulz KF, Altman D; CONSORT Group (Consolidated Standards of Reporting Trials). The CONSORT statement: revised recommendations for improving the quality of reports of parallel-group randomized trials. JAMA. 2001 Apr 18;285(15):1987-91. doi: 10.1001/jama.285.15.1987. PMID 11308435
- [Background] Azziz R. Controversy in clinical endocrinology: diagnosis of polycystic ovarian syndrome: the Rotterdam criteria are premature. J Clin Endocrinol Metab. 2006 Mar;91(3):781-5. doi: 10.1210/jc.2005-2153. Epub 2006 Jan 17. PMID 16418211
- [Background] Lessey BA, Ilesanmi AO, Lessey MA, Riben M, Harris JE, Chwalisz K. Luminal and glandular endometrial epithelium express integrins differentially throughout the menstrual cycle: implications for implantation, contraception, and infertility. Am J Reprod Immunol. 1996 Mar;35(3):195-204. doi: 10.1111/j.1600-0897.1996.tb00031.x. PMID 8962647
- [Background] Lessey BA, Castelbaum AJ, Buck CA, Lei Y, Yowell CW, Sun J. Further characterization of endometrial integrins during the menstrual cycle and in pregnancy. Fertil Steril. 1994 Sep;62(3):497-506. PMID 8062944
- [Background] Dehbashi S, Vafaei H, Parsanezhad MD, Alborzi S. Time of initiation of clomiphene citrate and pregnancy rate in polycystic ovarian syndrome. Int J Gynaecol Obstet. 2006 Apr;93(1):44-8. doi: 10.1016/j.ijgo.2005.10.015. Epub 2006 Mar 10. PMID 16530767
- [Background] Bayar U, Tanriverdi HA, Barut A, Ayoglu F, Ozcan O, Kaya E. Letrozole vs. clomiphene citrate in patients with ovulatory infertility. Fertil Steril. 2006 Apr;85(4):1045-8. doi: 10.1016/j.fertnstert.2005.09.045. Epub 2006 Mar 9. PMID 16580393
- [Background] Lessey BA, Castelbaum AJ, Sawin SW, Sun J. Integrins as markers of uterine receptivity in women with primary unexplained infertility. Fertil Steril. 1995 Mar;63(3):535-42. PMID 7851583
- [Background] Savaris RF, Pedrini JL, Flores R, Fabris G, Zettler CG. Expression of alpha 1 and beta 3 integrins subunits in the endometrium of patients with tubal phimosis or hydrosalpinx. Fertil Steril. 2006 Jan;85(1):188-92. doi: 10.1016/j.fertnstert.2005.06.039. PMID 16412752
- [Background] Hollis S, Campbell F. What is meant by intention to treat analysis? Survey of published randomised controlled trials. BMJ. 1999 Sep 11;319(7211):670-4. doi: 10.1136/bmj.319.7211.670. PMID 10480822
- [Derived] de Paula Guedes Neto E, Savaris RF, von Eye Corleta H, de Moraes GS, do Amaral Cristovam R, Lessey BA. Prospective, randomized comparison between raloxifene and clomiphene citrate for ovulation induction in polycystic ovary syndrome. Fertil Steril. 2011 Sep;96(3):769-73. doi: 10.1016/j.fertnstert.2011.06.067. Epub 2011 Jul 22. PMID 21782166

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between September 2008 and October 2009 at Hospital de Clínicas de Porto Alegre, a tertiary teaching hospital.
Pre-assignment Details: Women were excluded if they had elevated levels of thyroid-stimulating hormone, prolactin, or 17α-hydroxyprogesterone, if they had used oral contraceptives in the previous 2 months, or if they had a history of endometriosis.
Groups:
- Raloxiphene: Use of 100mg of raloxifene during days 5-9 of the menstrual cycle
Period: Overall Study
Arm/Group | Clomiphene | Raloxiphene
Started | 40 | 42
Completed | 37 | 31
Not Completed | 3 | 11
Not completed — Lost to Follow-up | 2 | 5
Not completed — no induction of menses | 1 | 4
Not completed — Pregnancy | 0 | 2

BASELINE CHARACTERISTICS:
Population: Numbers of participants for analysis was determined according to the sample size calculation
Groups:
- Total: Total of all reporting groups
Arm/Group | Raloxifene | Clomiphene | Total
Number analyzed (Participants) | 42 | 40 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 40 | 82
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.21 (5.3) | 28.7 (4.8) | 28.4 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 40 | 82
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 42 | 40 | 82

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Ovulation Detected by Ultrasound
Description: Ovulation detected by ultrasound was defined as the percentage of a participants with ovulation detected by ultrasound, defined as the dominant follicle and its subsequent collapse. If a dominant follicle was not observed by day 21 after menses, the ovulation induction was considered to be a failure.
Time Frame: cycle day 14-20
Population: intention to treat.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Clomiphene | Raloxifene
Number analyzed (Participants) | 40 | 42
percentage of participants | 52.5 [36.1 to 68.5] | 40.4 [25.6 to 56.6]
Statistical Analysis 1: Comparison: Clomiphene vs Raloxifene; The null hypothesis is that there is no significant difference between two drugs for ovulation induction.A sample size of 40 women per arm was calculated for this superiority trial, considering an alpha and beta error of 0.05 and 0.2, respectively, to find an absolute difference of 30% in the ovulation rate between groups, based on a previous study published by Mitwally and Casper (18) where the ovulation rate with CC was approximately 45%; Test type: Superiority or Other; p = 0.3, Fisher Exact; Mean Difference (Final Values) = 12, 95% CI 2-sided [-9 to 33]

2. Secondary Outcome: Serum Levels of Progesterone
Description: The level of serum progesterone that indicated ovulation was considered to be 3 ng/mL or greater, on days 8 to 10 after ovulation.
Time Frame: 8-10 days after ovulation
Population: Intention to treat.Cases that were lost to follow-up observation, dropped out of the study, failed to collect progesterone on days 22 to 24, and lacked menses after medroxyprogesterone acetate treatment were considered as failures according to the intention-to-treat analysis.
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Clomiphene | Raloxiphene
Number analyzed (Participants) | 40 | 42
ng/mL | 26.1 [13.8 to 42] | 40 [24.8 to 56.6]
Statistical Analysis 1: Comparison: Clomiphene vs Raloxiphene; Null hypothesis: There is no difference between the mean values of progesterone between both groups; Test type: Superiority or Other; p = 0.2, t-test, 2 sided; Mean Difference (Final Values) = 13, 95% CI 2-sided [-6 to 34]

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Clomiphene Citrate: Use of 100mg of clomiphene citrate during days 5-9 of the menstrual cycle
  clomiphene citrate: 100mg PO on days 5-9 of the menstrual cycle
  One woman in the CC group had nausea, headache, and abdominal bloating.
- Raloxifene: Use of 100mg of raloxifene during days 5-9 of the menstrual cycle
  raloxifene: 100mg PO on days 5-9 of the menstrual cycle
  Two cases: one woman had nausea, and the other woman had nausea, headache, and pelvic pain. All mild
Arm/Group | Clomiphene Citrate | Raloxifene
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/42
Other Adverse Events (participants affected / at risk) | 1/40 | 2/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clomiphene Citrate (N=40) | Raloxifene (N=42)
nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
headache (Nervous system disorders) | 1 (1) | 1 (1) — headache
abdominal bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No